CLINICAL TRIAL: NCT01217112
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Group, Pilot Study of 1:1 and 20:1 Ratio of Formulated GWP42003 : GWP42004 Plus GWP42003 and GWP42004 Alone in the Treatment of Dyslipidaemia in Subjects With Type 2 Diabetes
Brief Title: GWMD1092 - GWP42003 : GWP42004 Together Plus Alone in Type II Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWMD1092; 2010-020458-33 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Dyslipidemias; Diabetes Mellitus, Type 2
Keywords: Dyslipidemias; Diabetes; Liver Fat; Body Fat
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2; Diabetes Mellitus; Fatty Liver | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- GWP42004 and placebo (Active Comparator): Contains GWP42004 5 mg and placebo (excipients only)
  Interventions: Drug: GWP42004; Drug: Placebo
- 1:1 GWP42003 : GWP42004 (Active Comparator): Contains 5 mg each of GWP42003 and GWP42004
  Interventions: Drug: GWP42003; Drug: GWP42004
- 20:1 GWP42003 : GWP42004 (Active Comparator): Contains 100 mg GWP42003 and 5 mg GWP42004
  Interventions: Drug: GWP42003; Drug: GWP42004
- Placebo (Placebo Comparator): Contains excipients only
  Interventions: Drug: Placebo
- GWP42003 and placebo (Active Comparator): Contains 100 mg GWP42003 and placebo (excipients only)
  Interventions: Drug: GWP42003; Drug: Placebo

INTERVENTIONS:
Drug: GWP42003 — 100 mg capsules, PO, BD, 91 days
  Other Names: Cannabidiol; CBD
  Arms: 20:1 GWP42003 : GWP42004; GWP42003 and placebo
Drug: GWP42003 — 5 mg capsules, PO, BD, 91 days
  Other Names: Cannabidiol; CBD
  Arms: 1:1 GWP42003 : GWP42004
Drug: GWP42004 — 5 mg capsules, PO, BD, 91 days
  Other Names: delta-9-tetrahydrocannabivarin; THCV
  Arms: 1:1 GWP42003 : GWP42004; 20:1 GWP42003 : GWP42004; GWP42004 and placebo
Drug: Placebo — 0 mg capsules, QDS, PO, 91 days
  Arms: GWP42003 and placebo; GWP42004 and placebo; Placebo

SUMMARY:
This 15-19 week study is being conducted by GW Pharma Ltd as a pilot study in order to determine the efficacy and safety of two cannabinoids: GWP42004 and GWP42003 alone, or in combination in patients with Type 2 diabetes. This is the first study to determine whether the study medications have a positive benefit for subjects on their cholesterol levels, body weight, liver fat content and other metabolic parameters compared with a placebo medication.

DETAILED DESCRIPTION:
In this study there was a 1-5 week baseline period followed by a 13 week treatment period, and a one week follow-up. Eligible subjects entered the study at a screening visit (Visit 1) before returning for randomisation (Visit 2, Day 1). At the discretion of the investigator (based on individual subjects), Visit 1 could be split into two separate visits (Visits 1A and B) to allow a 21-day washout period of prohibited medications prior to blood sampling for eligibility. Further outpatient study visits (for assessment purposes) took place at the study site at the end of Week 4 of treatment (Visit 3, Day 29), and at the overall end of treatment at Week 13 (Visit 5, Day 92). A telephone assessment was also performed at Day 57 (Visit 4) and at Week 14 (Visit 6, Day 99) for safety follow-up purposes.

During the 13 week randomised treatment phase, subjects received blinded, oral doses of their allocated randomised treatment twice daily. Treatment was self-administered on an outpatient basis, once in the morning and once in the evening for 13 weeks. Subjects were instructed to time study medication to 30 minutes before breakfast and evening meals.

Physical and metabolic parameters were assessed before, during and after treatment to evaluate clinical response. Diabetic and dyslipidaemic medication usage (where applicable), and appetite 0-10 NRS data were collected daily during the treatment period, using the study diary.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Type 2 diabetes, with residual islet cell function;
* Diet controlled or receiving oral anti-diabetic treatment (metformin or other biguanides and/or sulphonyl ureas) who have received a stable dose for at least 3 months prior to enrollment;
* High Density Lipoprotein cholesterol ≤ 1.3mmol/L (females), ≤ 1.2mmol/L (males);
* Glycosylated haemoglobin levels of ≤ 10%;
* Triglycerides ≤ 10mmol/L;
* Willing to maintain a stable dose of oral anti-diabetic and/or lipid-lowering agents/medications that may have an effect on plasma/serum glucose, insulin or lipid parameters for the duration of the study, where applicable;
* No changes in diet or exercise for four weeks prior to and subject agrees to keep stable for the duration of the study (in the opinion of the investigator);

Exclusion Criteria:

* Subject is taking insulin (i.e. they are insulin-dependent);
* Taking the following categories of medicines: fibrates, Thiazolidinediones, therapeutic Omega-3 fatty acids, alpha-glucosidase inhibitors and unwilling abstain for the duration of the study;
* Currently using or has used recreational cannabis, medicinal cannabis, cannabinoid medications (including Sativex®), or synthetic cannabinoid based medications within 30 days prior to study entry and unwilling to abstain for the duration for the study;
* Any known or suspected history of:

  * alcohol or substance abuse
  * epilepsy or recurrent seizures;
* Any known or suspected history of depression sufficient to require treatment with antidepressants or disrupt ordinary life at the discretion of the investigator);
* Subject who has significant history of anxiety, suicidal ideation or self-harm;
* Clinically significant cardiac, renal or hepatic impairment in the opinion of the investigator;
* Genetic dyslipidaemic condition in the opinion of the investigator;
* Currently taking a lipid lowering agent and a stable dose has not been maintained for at least four weeks randomisation (Visit 2);
* Female subject, who is pregnant, lactating or planning pregnancy during the course of the study and for three months from date of last dose;
* Female subjects of child bearing potential unless willing to use two forms of contraception, one of which must be barrier contraception (e.g. female condom or occlusive cap (diaphragm or cervical vault/caps) with spermicide) during the study and for three months thereafter;
* Male subjects whose partner is of child bearing potential, unless willing to use an appropriate barrier method of contraception (condom and spermicide) in addition to having their female partner use another form of barrier contraception (e.g. female condom or occlusive cap (diaphragm or cervical vault/caps) with spermicide) during the study and for three months thereafter;
* Body weight > 150kg;
* Travel outside the country of residence planned during the study;
* Currently receiving a prohibited medication and unwilling to stop at the screening visit and for the duration of the study;
* Received an unapproved Investigational Medicinal Product (IMP) within the 30 days before the screening visit;
* In the opinion of the investigator, is not considered to be suitable for the study;
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP(s);
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study;
* Has a postural drop of ≥ 20 mmHg in systolic blood pressure at Visit 1;
* Any abnormalities identified during the physical exam at Visit 1 that in the opinion of the investigator, would prevent the subject from safe participation in the study;
* Unwilling to abstain from donation of blood during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Woolpit Health Centre, Bury Saint Edmonds
  - Mount Farm Surgery, Bury Saint Edmonds
  - University of Nottingham, Medical School at Derby, Royal Derby Hospital, Derby
  - James Paget University Hospital, Gorleston-on-Sea, Norfolk
  - MAC UK Neuroscience Ltd., Manchester

REFERENCES:
- [Derived] Jadoon KA, Ratcliffe SH, Barrett DA, Thomas EL, Stott C, Bell JD, O'Sullivan SE, Tan GD. Efficacy and Safety of Cannabidiol and Tetrahydrocannabivarin on Glycemic and Lipid Parameters in Patients With Type 2 Diabetes: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Pilot Study. Diabetes Care. 2016 Oct;39(10):1777-86. doi: 10.2337/dc16-0650. Epub 2016 Aug 29. PMID 27573936

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Started | 11 | 12 | 13 | 12 | 14
Completed | 11 | 10 | 12 | 10 | 13
Not Completed | 0 | 2 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 11 | 8 | 10 | 48
  >=65 years | 3 | 1 | 2 | 4 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.33 (8.75) | 57.96 (8.11) | 56.80 (9.92) | 62.45 (12.58) | 58.63 (7.72) | 58.98 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 2 | 7 | 20
  Male | 6 | 9 | 10 | 10 | 7 | 42
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 12 | 13 | 12 | 14 | 62

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Mean Serum High Density Lipoprotein Cholesterol Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum High Density Lipoprotein cholesterol. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: The analysis population comprised all randomised subjects who received at least one dose of study medication and had on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
mmol/l | 0.00 (0.09) | 0.04 (0.07) | -0.04 (0.14) | 0.00 (0.14) | 0.02 (0.09)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; Data was analysed by analysis of covariance (ANCOVA). The fitted ANCOVA models included the baseline parameter scores as covariate, with treatment group and gender as factors. All statistical tests were two-sided at the 10% significance level; Test type: Superiority or Other; p = 0.766, ANCOVA; Mean Difference (Final Values) = -0.01, 90% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; Data was analysed by ANCOVA. The fitted ANCOVA models included the baseline parameter scores as covariate, with treatment group and gender as factors. All statistical tests were two-sided at the 10% significance level; Test type: Superiority or Other; p = 0.424, ANCOVA; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.04 to 0.11], Standard Error of Mean 0.043
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.412, ANCOVA; Mean Difference (Final Values) = -0.03, 90% CI 2-sided [-0.10 to 0.04], Standard Error of Mean 0.041
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.668, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.05 to 0.09], Standard Error of Mean 0.043

2. Secondary Outcome: The Change From Baseline in Mean High Density Lipoprotein Cholesterol Concentration by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of High Density Lipoprotein cholesterol by ultracentrifugation. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
mmol/l | -0.04 (0.12) | -0.06 (0.08) | -0.11 (0.08) | -0.01 (0.16) | -0.02 (0.11)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.978, ANCOVA; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.08 to 0.08], Standard Error of Mean 0.046
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.864, ANCOVA; Mean Difference (Final Values) = -0.01, 90% CI 2-sided [-0.08 to 0.07], Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.537, ANCOVA; Mean Difference (Final Values) = -0.03, 90% CI 2-sided [-0.12 to 0.05], Standard Error of Mean 0.050
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.260, ANCOVA; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.02 to 0.13], Standard Error of Mean 0.045

3. Secondary Outcome: The Change From Baseline in Mean Serum Total Cholesterol Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum total cholesterol. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
mmol/l | -0.53 (0.78) | -0.27 (0.32) | -0.22 (0.50) | -0.13 (0.44) | -0.09 (0.39)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.088, ANCOVA; Mean Difference (Final Values) = -0.31, 90% CI 2-sided [-0.61 to -0.01], Standard Error of Mean 0.180
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.583, ANCOVA; Mean Difference (Final Values) = 0.10, 90% CI 2-sided [-0.20 to 0.39], Standard Error of Mean 0.177
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.388, ANCOVA; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [-0.14 to 0.43], Standard Error of Mean 0.169
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.580, ANCOVA; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.19 to 0.38], Standard Error of Mean 0.170

4. Secondary Outcome: The Change From Baseline in Mean Total Cholesterol Concentration by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum total cholesterol by ultracentrifugation. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
mmol/l | -0.12 (0.83) | -0.23 (0.28) | -0.11 (0.52) | -0.11 (0.45) | -0.16 (0.33)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.829, ANCOVA; Mean Difference (Final Values) = 0.04, 90% CI 2-sided [-0.29 to 0.37], Standard Error of Mean 0.198
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.575, ANCOVA; Mean Difference (Final Values) = 0.11, 90% CI 2-sided [-0.22 to 0.44], Standard Error of Mean 0.196
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.356, ANCOVA; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.15 to 0.53], Standard Error of Mean 0.203
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.472, ANCOVA; Mean Difference (Final Values) = 0.14, 90% CI 2-sided [-0.18 to 0.45], Standard Error of Mean 0.188

5. Secondary Outcome: The Change From Baseline in Mean Serum Low Density Lipoprotein Cholesterol Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum Low Density Lipoprotein cholesterol. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 8 | 11 | 11 | 12 | 13
mmol/l | -0.29 (0.62) | -0.13 (0.36) | -0.11 (0.40) | -0.02 (0.50) | 0.07 (0.33)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.115, ANCOVA; Mean Difference (Final Values) = -0.29, 90% CI 2-sided [-0.59 to 0.01], Standard Error of Mean 0.181
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.782, ANCOVA; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.25 to 0.35], Standard Error of Mean 0.177
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.902, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.27 to 0.31], Standard Error of Mean 0.173
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.993, ANCOVA; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.28 to 0.28], Standard Error of Mean 0.166

6. Secondary Outcome: The Change From Baseline in Mean Low Density Lipoprotein Cholesterol Concentration by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of Low Density Lipoprotein cholesterol by ultracentrifugation. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
mmol/l | -0.03 (0.49) | -0.16 (0.26) | -0.08 (0.43) | -0.08 (0.41) | -0.06 (0.19)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.956, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.23 to 0.25], Standard Error of Mean 0.143
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.705, ANCOVA; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.19 to 0.30], Standard Error of Mean 0.144
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.466, ANCOVA; Mean Difference (Final Values) = 0.11, 90% CI 2-sided [-0.14 to 0.36], Standard Error of Mean 0.148
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.876, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.21 to 0.25], Standard Error of Mean 0.136

7. Secondary Outcome: The Change From Baseline in Mean Serum High Density Lipoprotein : Low Density Lipoprotein Cholesterol Ratio After 91 Days (13 Weeks) of Treatment
Description: An increase from baseline (i.e. a positive value) to the end of treatment in the High Density Lipoprotein : Low Density Lipoprotein cholesterol ratio indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 8 | 11 | 11 | 12 | 13
ratio | 0.03 (0.11) | 0.04 (0.05) | -0.02 (0.08) | 0.02 (0.09) | 0.01 (0.06)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.408, ANCOVA; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.03 to 0.09], Standard Error of Mean 0.034
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.714, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.04 to 0.07], Standard Error of Mean 0.032
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.267, ANCOVA; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-0.09 to 0.02], Standard Error of Mean 0.032
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.484, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.03 to 0.08], Standard Error of Mean 0.032

8. Secondary Outcome: The Change From Baseline in Mean High Density Lipoprotein : Low Density Lipoprotein Cholesterol Ratio by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: as for outcome 7
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
ratio | -0.01 (0.11) | 0.00 (0.05) | -0.02 (0.08) | 0.03 (0.12) | 0.01 (0.06)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.560, ANCOVA; Mean Difference (Final Values) = -0.02, 90% CI 2-sided [-0.09 to 0.04], Standard Error of Mean 0.039
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.956, ANCOVA; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.06 to 0.06], Standard Error of Mean 0.037
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.403, ANCOVA; Mean Difference (Final Values) = -0.03, 90% CI 2-sided [-0.10 to 0.03], Standard Error of Mean 0.039
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.617, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.04 to 0.08], Standard Error of Mean 0.037

9. Secondary Outcome: The Change From Baseline in Mean Very Low Density Lipoprotein Cholesterol Concentration by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of Very Low Density Lipoprotein cholesterol by ultracentrifugation. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
mmol/l | -0.06 (0.37) | -0.01 (0.16) | 0.08 (0.19) | -0.02 (0.24) | -0.08 (0.31)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.815, ANCOVA; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.16 to 0.21], Standard Error of Mean 0.108
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.418, ANCOVA; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.09 to 0.26], Standard Error of Mean 0.105
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.236, ANCOVA; Mean Difference (Final Values) = 0.13, 90% CI 2-sided [-0.05 to 0.32], Standard Error of Mean 0.111
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.556, ANCOVA; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.11 to 0.23], Standard Error of Mean 0.103

10. Secondary Outcome: The Change From Baseline in Mean Serum Triglyceride Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum triglyceride concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
mmol/l | -0.47 (0.54) | 0.14 (0.28) | 0.09 (0.55) | 0.09 (0.66) | -0.12 (0.80)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.329, ANCOVA; Mean Difference (Final Values) = -0.24, 90% CI 2-sided [-0.64 to 0.17], Standard Error of Mean 0.241
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.232, ANCOVA; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-0.11 to 0.68], Standard Error of Mean 0.236
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.164, ANCOVA; Mean Difference (Final Values) = 0.31, 90% CI 2-sided [-0.06 to 0.68], Standard Error of Mean 0.222
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.302, ANCOVA; Mean Difference (Final Values) = 0.24, 90% CI 2-sided [-0.15 to 0.63], Standard Error of Mean 0.232

11. Secondary Outcome: The Change From Baseline in Mean Triglyceride Concentration by Ultracentrifugation After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of triglyceride concentrations by ultracentrifugation. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 9 | 12 | 14
mmol/l | -0.16 (0.56) | 0.12 (0.26) | 0.16 (0.34) | 0.05 (0.59) | -0.03 (0.74)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.614, ANCOVA; Mean Difference (Final Values) = -0.12, 90% CI 2-sided [-0.50 to 0.27], Standard Error of Mean 0.231
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.669, ANCOVA; Mean Difference (Final Values) = 0.10, 90% CI 2-sided [-0.28 to 0.48], Standard Error of Mean 0.227
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.621, ANCOVA; Mean Difference (Final Values) = 0.12, 90% CI 2-sided [-0.28 to 0.52], Standard Error of Mean 0.240
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.867, ANCOVA; Mean Difference (Final Values) = 0.04, 90% CI 2-sided [-0.33 to 0.41], Standard Error of Mean 0.222

12. Secondary Outcome: The Change From Baseline in Mean Serum Apolipoprotein A Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum Apolipoprotein A. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 14
umol/l | -2.86 (8.84) | -3.51 (10.88) | -4.92 (6.04) | 0.64 (11.32) | -3.41 (6.22)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.335, ANCOVA; Mean Difference (Final Values) = 2.55, 90% CI 2-sided [-1.84 to 6.95], Standard Error of Mean 2.624
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.358, ANCOVA; Mean Difference (Final Values) = 2.36, 90% CI 2-sided [-1.90 to 6.62], Standard Error of Mean 2.545
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.900, ANCOVA; Mean Difference (Final Values) = 0.30, 90% CI 2-sided [-3.72 to 4.33], Standard Error of Mean 2.406
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Final Values) = 6.02, 90% CI 2-sided [1.86 to 10.19], Standard Error of Mean 2.486

13. Secondary Outcome: The Change From Baseline in Mean Serum Apolipoprotein B Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum Apolipoprotein B. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
umol/l | -0.19 (0.84) | 0.18 (0.51) | 0.11 (0.53) | 0.08 (0.66) | 0.16 (0.42)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.325, ANCOVA; Mean Difference (Final Values) = -0.24, 90% CI 2-sided [-0.65 to 0.17], Standard Error of Mean 0.245
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.438, ANCOVA; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.21 to 0.59], Standard Error of Mean 0.238
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.701, ANCOVA; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.29 to 0.47], Standard Error of Mean 0.226
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.624, ANCOVA; Mean Difference (Final Values) = -0.11, 90% CI 2-sided [-0.50 to 0.27], Standard Error of Mean 0.232

14. Secondary Outcome: The Change From Baseline in Mean Serum Apolipoprotein B : Apolipoprotein A Ratio After 91 Days (13 Weeks) of Treatment
Description: A decrease from baseline to the end of treatment (i.e. a negative value) in the Apolipoprotein B : Apolipoprotein A ratio indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
ratio | -0.01 (0.23) | 0.07 (0.15) | 0.08 (0.13) | 0.01 (0.14) | 0.07 (0.12)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.233, ANCOVA; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.17 to 0.03], Standard Error of Mean 0.058
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.727, ANCOVA; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.07 to 0.11], Standard Error of Mean 0.056
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.593, ANCOVA; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.06 to 0.12], Standard Error of Mean 0.053
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.075, ANCOVA; Mean Difference (Final Values) = -0.10, 90% CI 2-sided [-0.20 to -0.01], Standard Error of Mean 0.056

15. Secondary Outcome: The Change From Baseline in Mean Serum Non-Esterified Fatty Acid Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of serum Non-Esterified Fatty Acid concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 13
mmol/l | 0.06 (0.17) | -0.03 (0.23) | -0.05 (0.30) | -0.02 (0.18) | 0.01 (0.15)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.236, ANCOVA; Mean Difference (Final Values) = 0.10, 90% CI 2-sided [-0.04 to 0.24], Standard Error of Mean 0.084
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.579, ANCOVA; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.09 to 0.18], Standard Error of Mean 0.082
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.837, ANCOVA; Mean Difference (Final Values) = -0.02, 90% CI 2-sided [-0.15 to 0.11], Standard Error of Mean 0.077
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.467, ANCOVA; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.08 to 0.19], Standard Error of Mean 0.081

16. Secondary Outcome: The Change From Baseline in Mean Fasting Glucose Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of fasting glucose concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 11 | 13
mmol/l | -0.23 (2.02) | 0.44 (2.00) | 0.41 (0.82) | -0.76 (1.00) | 0.38 (1.15)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.533, ANCOVA; Mean Difference (Final Values) = -0.38, 90% CI 2-sided [-1.41 to 0.64], Standard Error of Mean 0.613
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.804, ANCOVA; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [-0.84 to 1.13], Standard Error of Mean 0.585
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.916, ANCOVA; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.87 to 0.99], Standard Error of Mean 0.556
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.040, ANCOVA; Mean Difference (Final Values) = -1.23, 90% CI 2-sided [-2.20 to -0.25], Standard Error of Mean 0.583

17. Secondary Outcome: The Change From Baseline in Mean Fructosamine Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of fructosamine concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 10 | 13 | 12 | 13
umol/l | 2.8 (42.06) | 14.5 (29.53) | -2.6 (20.41) | 1.1 (11.68) | 9.5 (19.68)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.366, ANCOVA; Mean Difference (Final Values) = -9.90, 90% CI 2-sided [-28.06 to 8.27], Standard Error of Mean 10.838
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.844, ANCOVA; Mean Difference (Final Values) = 2.11, 90% CI 2-sided [-15.81 to 20.03], Standard Error of Mean 10.692
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.118, ANCOVA; Mean Difference (Final Values) = -15.96, 90% CI 2-sided [-32.76 to 0.84], Standard Error of Mean 10.026
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.518, ANCOVA; Mean Difference (Final Values) = -6.67, 90% CI 2-sided [-23.86 to 10.51], Standard Error of Mean 10.256

18. Secondary Outcome: The Change From Baseline in Mean Glycated Haemoglobin Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of glycated haemoglobin concentrations. At both time points, values were calculated as a percentage of total haemoglobin. A decrease from baseline to the end of treatment in base per cent values, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 12 | 14
percent | 0.14 (1.41) | 0.16 (0.44) | 0.08 (0.44) | -0.03 (0.22) | 0.31 (0.54)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.576, ANCOVA; Mean Difference (Final Values) = -0.17, 90% CI 2-sided [-0.66 to 0.33], Standard Error of Mean 0.294
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.648, ANCOVA; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-0.60 to 0.34], Standard Error of Mean 0.283
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.447, ANCOVA; Mean Difference (Final Values) = -0.21, 90% CI 2-sided [-0.66 to 0.24], Standard Error of Mean 0.269
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.273, ANCOVA; Mean Difference (Final Values) = -0.31, 90% CI 2-sided [-0.79 to 0.16], Standard Error of Mean 0.283

19. Secondary Outcome: The Change From Baseline to the End of 91 Days (13 Weeks) of Treatment in the Mean Serum Glucose Concentration Two Hours Post Glucose Challenge (Oral Glucose Tolerance Test [OGTT])
Description: A two-hour OGTT was performed to investigate the rate of glucose metabolism or clearance from the blood with treatment. Blood samples were taken at -15 and 0 minutes prior to a glucose drink and at 30, 60, 90, 120 and 180 minutes post drink. The OGTT measured the change from baseline in serum glucose levels at two hours (120 minutes) compared to 0 minutes. The extent of the elevation in blood glucose levels following a glucose drink were compared between baseline and the end of treatment. A reduction in the elevation of serum glucose levels at the end of treatment (i.e. a negative value) indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 6 | 10 | 12 | 11 | 13
mmol/l | -0.07 (1.89) | 1.09 (3.81) | -0.78 (1.51) | 0.22 (1.85) | 0.42 (1.44)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.615, ANCOVA; Mean Difference (Final Values) = -0.56, 90% CI 2-sided [-2.40 to 1.29], Standard Error of Mean 1.097
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.342, ANCOVA; Mean Difference (Final Values) = 0.93, 90% CI 2-sided [-0.70 to 2.57], Standard Error of Mean 0.973
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.314, ANCOVA; Mean Difference (Final Values) = -0.95, 90% CI 2-sided [-2.52 to 0.62], Standard Error of Mean 0.934
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.889, ANCOVA; Mean Difference (Final Values) = 0.14, 90% CI 2-sided [-1.48 to 1.75], Standard Error of Mean 0.964

20. Secondary Outcome: The Change From Baseline to the End of 91 Days (13 Weeks) of Treatment in the Mean Serum Insulin Concentration Two Hours Post Glucose Challenge (Oral Glucose Tolerance Test)
Description: At baseline and the end of treatment, blood samples were taken at -15 and 0 minutes prior to a glucose drink and at 30, 60, 90, 120 and 180 minutes post drink. The OGTT measured the change from baseline in serum insulin levels at two hours (120 minutes) compared to 0 minutes. The extent of the elevation in blood glucose levels following a glucose drink were compared between baseline and the end of treatment. An increase in the elevation of serum insulin levels from baseline to the end of treatment (i.e. a positive value) indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 9 | 12 | 11 | 13
pmol/l | 80.9 (223.91) | -156.6 (358.53) | -193.5 (232.17) | 83.5 (427.94) | -40.8 (475.88)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.764, ANCOVA; Mean Difference (Final Values) = 50.89, 90% CI 2-sided [-232.02 to 333.80], Standard Error of Mean 168.459
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.654, ANCOVA; Mean Difference (Final Values) = -70.76, 90% CI 2-sided [-333.96 to 192.44], Standard Error of Mean 156.720
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.450, ANCOVA; Mean Difference (Final Values) = -111.50, 90% CI 2-sided [-357.17 to 134.16], Standard Error of Mean 146.276
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.517, ANCOVA; Mean Difference (Final Values) = 97.42, 90% CI 2-sided [-153.02 to 347.86], Standard Error of Mean 149.124

21. Secondary Outcome: The Change From Baseline in Mean Fasting Insulin Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of fasting insulin concentrations. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 11 | 13
pmol/l | 12.01 (56.22) | -6.06 (104.78) | 13.44 (49.03) | 45.62 (183.92) | 2.79 (61.44)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.840, ANCOVA; Mean Difference (Final Values) = 8.33, 90% CI 2-sided [-60.28 to 76.94], Standard Error of Mean 40.940
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.834, ANCOVA; Mean Difference (Final Values) = 8.31, 90% CI 2-sided [-57.92 to 74.55], Standard Error of Mean 39.521
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.767, ANCOVA; Mean Difference (Final Values) = -11.62, 90% CI 2-sided [-77.06 to 53.81], Standard Error of Mean 39.044
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.289, ANCOVA; Mean Difference (Final Values) = 42.51, 90% CI 2-sided [-23.99 to 109.01], Standard Error of Mean 39.680

22. Secondary Outcome: The Change From Baseline in Mean C-peptide Concentration After 91 Days (13 Weeks) of Treatment
Description: At baseline and the end of treatment, an approximately 30 mL fasting blood sample was taken for measurement of C-peptide concentrations. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 12 | 12 | 14
nmol/l | 0.02 (0.15) | 0.09 (0.28) | -0.03 (0.18) | 0.12 (0.31) | 0.09 (0.25)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.569, ANCOVA; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-0.24 to 0.12], Standard Error of Mean 0.106
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.984, ANCOVA; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.17 to 0.17], Standard Error of Mean 0.101
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; v Data was analysed by ANCOVA. The fitted ANCOVA models included the baseline parameter scores as covariate, with treatment group and gender as factors. All statistical tests were two-sided at the 10% significance level; Test type: Superiority or Other; p = 0.176, ANCOVA; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-0.30 to 0.03], Standard Error of Mean 0.098
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.895, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.15 to 0.18], Standard Error of Mean 0.099

23. Secondary Outcome: The Change From Baseline in Mean Insulin Resistance Measured by Homeostasis Model Assessment 2 (HOMA2-IR) After 91 Days (13 Weeks) of Treatment
Description: Changes from baseline to the end of treatment in mean insulin resistance were calculated by HOMA2-IR. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin resistance, which is the reciprocal of insulin sensitivity (%S)(100/%S) as a percentage of a normal reference population (normal young adults). A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IR score
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 11 | 13
IR score | 0.19 (1.00) | -0.19 (2.54) | 0.35 (1.20) | 0.64 (3.15) | 0.09 (1.22)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.871, ANCOVA; Mean Difference (Final Values) = 0.12, 90% CI 2-sided [-1.13 to 1.37], Standard Error of Mean 0.745
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.826, ANCOVA; Mean Difference (Final Values) = 0.16, 90% CI 2-sided [-1.05 to 1.37], Standard Error of Mean 0.721
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.693, ANCOVA; Mean Difference (Final Values) = -0.28, 90% CI 2-sided [-1.46 to 0.90], Standard Error of Mean 0.703
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.536, ANCOVA; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [-0.76 to 1.66], Standard Error of Mean 0.722

24. Secondary Outcome: The Change From Baseline in Mean Insulin Sensitivity Measured by Homeostasis Model Assessment 2 (HOMA2) After 91 Days (13 Weeks) of Treatment
Description: Changes from baseline to the end of treatment in mean insulin sensitivity were calculated by HOMA2. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S) as a percentage of a normal reference population (normal young adults). An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent sensitivity
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 11 | 13
percent sensitivity | -5.26 (8.62) | -1.71 (12.62) | 1.71 (26.48) | 6.47 (27.00) | -4.07 (13.16)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.878, ANCOVA; Mean Difference (Final Values) = -1.33, 90% CI 2-sided [-15.80 to 13.13], Standard Error of Mean 8.633
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.919, ANCOVA; Mean Difference (Final Values) = 0.85, 90% CI 2-sided [-13.18 to 14.89], Standard Error of Mean 8.377
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.557, ANCOVA; Mean Difference (Final Values) = 4.72, 90% CI 2-sided [-8.67 to 18.11], Standard Error of Mean 7.989
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.275, ANCOVA; Mean Difference (Final Values) = 9.20, 90% CI 2-sided [-4.76 to 23.16], Standard Error of Mean 8.328

25. Secondary Outcome: The Change From Baseline in Mean Insulin B Cell Function Measured by Homeostasis Model Assessment 2 (HOMA2) After 91 Days (13 Weeks) of Treatment
Description: Changes from baseline to the end of treatment in mean insulin B Cell Function were calculated by HOMA2. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate beta cell function (%B) as a percentage of a normal reference population (normal young adults). An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent beta function
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 9 | 11 | 13 | 11 | 13
percent beta function | 8.13 (23.56) | -7.64 (35.00) | -1.31 (19.06) | 36.59 (70.55) | -2.41 (19.96)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.528, ANCOVA; Mean Difference (Final Values) = 10.45, 90% CI 2-sided [-17.12 to 38.01], Standard Error of Mean 16.445
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.990, ANCOVA; Mean Difference (Final Values) = 0.20, 90% CI 2-sided [-26.32 to 26.72], Standard Error of Mean 15.825
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.776, ANCOVA; Mean Difference (Final Values) = 4.39, 90% CI 2-sided [-21.37 to 30.15], Standard Error of Mean 15.369
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = 44.51, 90% CI 2-sided [17.98 to 71.05], Standard Error of Mean 15.834

26. Secondary Outcome: The Change From Baseline in Mean Body Mass Index After 91 Days (13 Weeks) of Treatment
Description: Body Mass Index was calculated at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
kg/m^2 | -0.38 (0.65) | -0.02 (0.72) | -0.20 (1.16) | -0.21 (1.09) | -0.50 (2.12)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.717, ANCOVA; Mean Difference (Final Values) = 0.20, 90% CI 2-sided [-0.70 to 1.09], Standard Error of Mean 0.536
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.218, ANCOVA; Mean Difference (Final Values) = 0.66, 90% CI 2-sided [-0.23 to 1.55], Standard Error of Mean 0.531
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.378, ANCOVA; Mean Difference (Final Values) = 0.46, 90% CI 2-sided [-0.40 to 1.32], Standard Error of Mean 0.514
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.361, ANCOVA; Mean Difference (Final Values) = 0.49, 90% CI 2-sided [-0.40 to 1.38], Standard Error of Mean 0.532

27. Secondary Outcome: The Change From Baseline in Mean Waist-to-hip Ratio After 91 Days (13 Weeks) of Treatment
Description: Subject's waist-to-hip ratios were calculated at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
ratio | -0.00 (0.06) | -0.00 (0.04) | 0.00 (0.03) | -0.00 (0.02) | -0.01 (0.02)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.417, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.01 to 0.03], Standard Error of Mean 0.013
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.340, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.01 to 0.04], Standard Error of Mean 0.013
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.915, ANCOVA; Mean Difference (Final Values) = -0.00, 90% CI 2-sided [-0.02 to 0.02], Standard Error of Mean 0.013
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.465, ANCOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.01 to 0.03], Standard Error of Mean 0.013

28. Secondary Outcome: The Change From Baseline in Mean Body Weight After 91 Days (13 Weeks) of Treatment
Description: Subject's body weights were measured at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
kg | -1.05 (1.88) | -0.10 (2.07) | -0.46 (3.40) | -0.66 (3.09) | -1.64 (6.66)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.646, ANCOVA; Mean Difference (Final Values) = 0.75, 90% CI 2-sided [-1.96 to 3.45], Standard Error of Mean 1.616
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.219, ANCOVA; Mean Difference (Final Values) = 1.99, 90% CI 2-sided [-0.69 to 4.66], Standard Error of Mean 1.598
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.307, ANCOVA; Mean Difference (Final Values) = 1.61, 90% CI 2-sided [-1.00 to 4.23], Standard Error of Mean 1.563
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.348, ANCOVA; Mean Difference (Final Values) = 1.52, 90% CI 2-sided [-1.17 to 4.22], Standard Error of Mean 1.612

29. Secondary Outcome: The Change From Baseline in Mean Waist Measurement After 91 Days (13 Weeks) of Treatment
Description: Subjects' waist measurements were taken at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
cm | 0.82 (3.90) | -0.17 (2.59) | 0.31 (4.31) | -0.39 (1.48) | -0.86 (2.55)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.187, ANCOVA; Mean Difference (Final Values) = 1.74, 90% CI 2-sided [-0.44 to 3.91], Standard Error of Mean 1.299
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.578, ANCOVA; Mean Difference (Final Values) = 0.72, 90% CI 2-sided [-1.43 to 2.86], Standard Error of Mean 1.280
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.368, ANCOVA; Mean Difference (Final Values) = 1.13, 90% CI 2-sided [-0.96 to 3.22], Standard Error of Mean 1.249
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.696, ANCOVA; Mean Difference (Final Values) = 0.51, 90% CI 2-sided [-1.67 to 2.69], Standard Error of Mean 1.304

30. Secondary Outcome: The Change From Baseline in Mean Hip Measurement After 91 Days (13 Weeks) of Treatment
Description: Subjects' hip measurements were taken at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
cm | 1.12 (4.93) | 0.07 (2.54) | 0.38 (3.48) | -0.19 (1.30) | -0.20 (2.86)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.327, ANCOVA; Mean Difference (Final Values) = 1.30, 90% CI 2-sided [-0.90 to 3.51], Standard Error of Mean 1.320
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.851, ANCOVA; Mean Difference (Final Values) = 0.25, 90% CI 2-sided [-1.93 to 2.43], Standard Error of Mean 1.303
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.672, ANCOVA; Mean Difference (Final Values) = 0.54, 90% CI 2-sided [-1.60 to 2.69], Standard Error of Mean 1.281
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.978, ANCOVA; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-2.26 to 2.18], Standard Error of Mean 1.327

31. Secondary Outcome: The Change From Baseline in Mean Visceral Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Visceral Abdominal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scans were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 11 | 12
litres | 0.10 (0.96) | 0.62 (1.02) | 0.42 (0.87) | -0.11 (0.78) | 0.27 (1.97)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.857, ANCOVA; Mean Difference (Final Values) = -0.09, 90% CI 2-sided [-0.95 to 0.76], Standard Error of Mean 0.512
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.543, ANCOVA; Mean Difference (Final Values) = 0.34, 90% CI 2-sided [-0.58 to 1.26], Standard Error of Mean 0.549
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.859, ANCOVA; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.74 to 0.92], Standard Error of Mean 0.495
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.467, ANCOVA; Mean Difference (Final Values) = -0.39, 90% CI 2-sided [-1.27 to 0.50], Standard Error of Mean 0.526

32. Secondary Outcome: The Change From Baseline in Mean Subcutaneous Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Subcutaneous Abdominal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scans were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 11 | 12
litres | -0.3 (1.05) | 0.5 (0.56) | -0.0 (0.66) | 0.1 (0.84) | 0.3 (1.39)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.124, ANCOVA; Mean Difference (Final Values) = -0.64, 90% CI 2-sided [-1.32 to 0.05], Standard Error of Mean 0.406
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.909, ANCOVA; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.68 to 0.79], Standard Error of Mean 0.439
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.245, ANCOVA; Mean Difference (Final Values) = -0.46, 90% CI 2-sided [-1.12 to 0.20], Standard Error of Mean 0.392
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.382, ANCOVA; Mean Difference (Final Values) = -0.36, 90% CI 2-sided [-1.05 to 0.33], Standard Error of Mean 0.412

33. Secondary Outcome: The Change From Baseline in Mean Total Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Total Abdominal Fat was measured by magnetic resonance imaging, and the results of the scans were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 11 | 12
litres | -0.23 (1.53) | 1.08 (1.42) | 0.37 (1.25) | -0.05 (1.52) | 0.59 (3.24)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.376, ANCOVA; Mean Difference (Final Values) = -0.75, 90% CI 2-sided [-2.15 to 0.66], Standard Error of Mean 0.837
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.688, ANCOVA; Mean Difference (Final Values) = 0.37, 90% CI 2-sided [-1.15 to 1.89], Standard Error of Mean 0.908
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.637, ANCOVA; Mean Difference (Final Values) = -0.38, 90% CI 2-sided [-1.73 to 0.96], Standard Error of Mean 0.803
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.355, ANCOVA; Mean Difference (Final Values) = -0.79, 90% CI 2-sided [-2.22 to 0.63], Standard Error of Mean 0.849

34. Secondary Outcome: The Change From Baseline in Mean Internal Non-Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Internal Non-Abdominal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | -0.22 (1.13) | -0.75 (0.87) | 0.02 (0.62) | -0.29 (0.75) | -0.37 (0.43)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.482, ANCOVA; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-0.39 to 0.95], Standard Error of Mean 0.391
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.708, ANCOVA; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.65 to 1.02], Standard Error of Mean 0.489
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.166, ANCOVA; Mean Difference (Final Values) = 0.62, 90% CI 2-sided [-0.12 to 1.37], Standard Error of Mean 0.434
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.424, ANCOVA; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [-0.37 to 1.03], Standard Error of Mean 0.408

35. Secondary Outcome: The Change From Baseline in Mean Subcutaneous Non-Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Subcutaneous Non-Abdominal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | 0.6 (2.98) | 0.4 (1.35) | 0.2 (1.37) | 0.8 (3.17) | -2.4 (2.45)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.022, ANCOVA; Mean Difference (Final Values) = 3.10, 90% CI 2-sided [0.94 to 5.25], Standard Error of Mean 1.260
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Final Values) = 4.07, 90% CI 2-sided [1.44 to 6.69], Standard Error of Mean 1.532
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.053, ANCOVA; Mean Difference (Final Values) = 2.85, 90% CI 2-sided [0.45 to 5.25], Standard Error of Mean 1.400
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.012, ANCOVA; Mean Difference (Final Values) = 3.56, 90% CI 2-sided [1.33 to 5.78], Standard Error of Mean 1.299

36. Secondary Outcome: The Change From Baseline in Mean Total Non-Abdominal Fat After 91 Days (13 Weeks) of Treatment
Description: Total Non-Abdominal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | 0.33 (3.81) | -0.36 (1.52) | 0.18 (1.99) | 0.56 (3.87) | -2.81 (2.37)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.032, ANCOVA; Mean Difference (Final Values) = 3.35, 90% CI 2-sided [0.84 to 5.85], Standard Error of Mean 1.463
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.026, ANCOVA; Mean Difference (Final Values) = 4.27, 90% CI 2-sided [1.18 to 7.35], Standard Error of Mean 1.798
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.046, ANCOVA; Mean Difference (Final Values) = 3.44, 90% CI 2-sided [0.65 to 6.22], Standard Error of Mean 1.626
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.018, ANCOVA; Mean Difference (Final Values) = 3.86, 90% CI 2-sided [1.26 to 6.45], Standard Error of Mean 1.512

37. Secondary Outcome: The Change From Baseline in Mean Total Internal Fat After 91 Days (13 Weeks) of Treatment
Description: Total Internal Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | -0.09 (2.13) | 0.46 (0.56) | 0.40 (1.07) | -0.52 (1.29) | -0.88 (1.36)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.294, ANCOVA; Mean Difference (Final Values) = 0.87, 90% CI 2-sided [-0.52 to 2.25], Standard Error of Mean 0.806
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.092, ANCOVA; Mean Difference (Final Values) = 1.74, 90% CI 2-sided [0.05 to 3.43], Standard Error of Mean 0.988
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.173, ANCOVA; Mean Difference (Final Values) = 1.26, 90% CI 2-sided [-0.28 to 2.79], Standard Error of Mean 0.893
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.545, ANCOVA; Mean Difference (Final Values) = 0.51, 90% CI 2-sided [-0.92 to 1.95], Standard Error of Mean 0.837

38. Secondary Outcome: The Change From Baseline in Mean Total Subcutaneous Fat After 91 Days (13 Weeks) of Treatment
Description: Total Subcutaneous Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | 0.22 (2.63) | 1.11 (0.78) | 0.01 (1.88) | 1.08 (3.26) | -2.44 (2.25)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.038, ANCOVA; Mean Difference (Final Values) = 2.67, 90% CI 2-sided [0.59 to 4.75], Standard Error of Mean 1.214
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 4.71, 90% CI 2-sided [2.16 to 7.26], Standard Error of Mean 1.486
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.088, ANCOVA; Mean Difference (Final Values) = 2.40, 90% CI 2-sided [0.09 to 4.72], Standard Error of Mean 1.350
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Final Values) = 3.54, 90% CI 2-sided [1.39 to 5.68], Standard Error of Mean 1.252

39. Secondary Outcome: The Change From Baseline in Mean Total Fat After 91 Days (13 Weeks) of Treatment
Description: Total Fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | 0.13 (4.61) | 1.57 (0.46) | 0.40 (2.65) | 0.57 (4.34) | -3.31 (2.91)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.064, ANCOVA; Mean Difference (Final Values) = 3.53, 90% CI 2-sided [0.42 to 6.64], Standard Error of Mean 1.814
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = 6.55, 90% CI 2-sided [2.72 to 10.38], Standard Error of Mean 2.237
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.084, ANCOVA; Mean Difference (Final Values) = 3.65, 90% CI 2-sided [0.19 to 7.10], Standard Error of Mean 2.016
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.041, ANCOVA; Mean Difference (Final Values) = 4.05, 90% CI 2-sided [0.84 to 7.25], Standard Error of Mean 1.871

40. Secondary Outcome: The Change From Baseline in Mean Abdominal Adiposity After 91 Days (13 Weeks) of Treatment
Description: Abdominal Adiposity was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 7 | 4 | 6 | 6 | 7
litres | -0.02 (0.08) | 0.05 (0.06) | -0.01 (0.06) | 0.01 (0.08) | 0.04 (0.10)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.129, ANCOVA; Mean Difference (Net) = -0.07, 90% CI 2-sided [-0.14 to 0.01], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.961, ANCOVA; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.08 to 0.09], Standard Error of Mean 0.051
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.128, ANCOVA; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.16 to 0.01], Standard Error of Mean 0.048
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.300, ANCOVA; Mean Difference (Final Values) = -0.05, 90% CI 2-sided [-0.12 to 0.03], Standard Error of Mean 0.045

41. Secondary Outcome: The Change From Baseline in Mean % Liver Fat After 91 Days (13 Weeks) of Treatment
Description: Percentage liver fat was measured by magnetic resonance imaging at baseline and the end of treatment, and the results of the scan were analysed blind by a single independent reviewer. A decrease from baseline to the end of treatment in base per cent values, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent liver fat
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 11 | 11
percent liver fat | -1.12 (19.75) | 0.37 (7.15) | -4.73 (9.87) | 0.77 (10.56) | -2.95 (12.40)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.625, ANCOVA; Mean Difference (Final Values) = 2.65, 90% CI 2-sided [-6.37 to 11.67], Standard Error of Mean 5.380
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.226, ANCOVA; Mean Difference (Final Values) = 6.77, 90% CI 2-sided [-2.48 to 16.02], Standard Error of Mean 5.519
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.904, ANCOVA; Mean Difference (Final Values) = 0.62, 90% CI 2-sided [-7.94 to 9.18], Standard Error of Mean 5.103
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.285, ANCOVA; Mean Difference (Final Values) = 6.17, 90% CI 2-sided [-3.41 to 15.75], Standard Error of Mean 5.710

42. Secondary Outcome: The Change From Baseline in Mean Appetite 0-10 Numerical Rating Scale Score After 91 Days (13 Weeks) of Treatment
Description: Subjects scored their appetite daily using an appetite 0-10 numerical rating scale score where 0 = no appetite (don't feel hungry) and 10 = maximum appetite (completely hungry all the time). The mean change from baseline to the end of treatment in scores were calculated. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Time Frame: Baseline (Day 1) and End of treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 10 | 12 | 13 | 11 | 14
units on a scale | -1.19 (2.02) | -0.84 (1.96) | -0.69 (0.99) | -0.36 (2.01) | -0.59 (1.10)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.138, ANCOVA; Mean Difference (Final Values) = -0.85, 90% CI 2-sided [-1.81 to 0.10], Standard Error of Mean 0.568
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.505, ANCOVA; Mean Difference (Final Values) = -0.37, 90% CI 2-sided [-1.28 to 0.55], Standard Error of Mean 0.547
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.743, ANCOVA; Mean Difference (Final Values) = 0.18, 90% CI 2-sided [-0.73 to 1.08], Standard Error of Mean 0.540
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.540, ANCOVA; Mean Difference (Final Values) = 0.35, 90% CI 2-sided [-0.60 to 1.29], Standard Error of Mean 0.565

43. Secondary Outcome: Adverse Events as a Measure of Patient Safety
Description: The incidence of treatment-emergent adverse events was recorded for the study duration, and the number of patients who experienced an adverse event is presented.
Time Frame: Day 1 - Day 92
Population: All correctly randomised subjects who received at least one dose of study treatment were included and analysed according to the treatment received.
Measure: Number; unit: participants
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 14
participants | 7 | 8 | 11 | 11 | 13

44. Secondary Outcome: The Change From Baseline in Mean Beck Depression Inventory-II (BDI-II) Score at the End of 91 Days (13 Weeks) of Treatment
Description: The BDI-II is a 21 question, multiple choice, self-reported inventory, and is one of the most widely used instruments for measuring the severity of depression. The 21 questions or items each had four possible responses. Each response was assigned a score ranging from zero to three, indicating the severity of the symptom, with a total possible score ranging from zero to 63. A score between zero and 13 indicates 'minimal depression'. A score between 14 and 19 indicates 'mild depression'. A score between 20 and 28 indicates 'moderate depression', and a score between 29 and 63 indicates 'severe depression'. As such, an increase from baseline to the end of treatment, a positive value, indicates a deterioration.
Time Frame: Baseline (Day 1) and the End of Treatment (Day 92)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 12 | 13
units on a scale | 0.27 (1.27) | 4.91 (8.08) | 0.85 (2.23) | 0.58 (2.15) | -0.08 (4.17)
Statistical Analysis 1: Comparison: 1:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.701, ANCOVA; Mean Difference (Final Values) = 0.64, 90% CI 2-sided [-2.14 to 3.43], Standard Error of Mean 1.664
Statistical Analysis 2: Comparison: 20:1 GWP42003 : GWP42004 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = 4.77, 90% CI 2-sided [1.99 to 7.55], Standard Error of Mean 1.662
Statistical Analysis 3: Comparison: GWP42003 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.542, ANCOVA; Mean Difference (Final Values) = 0.98, 90% CI 2-sided [-1.68 to 3.64], Standard Error of Mean 1.589
Statistical Analysis 4: Comparison: GWP42004 and Placebo vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.827, ANCOVA; Mean Difference (Final Values) = 0.36, 90% CI 2-sided [-2.36 to 3.08], Standard Error of Mean 1.627

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the study (up to 133 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | 1:1 GWP42003 : GWP42004 | 20:1 GWP42003 : GWP42004 | GWP42003 and Placebo | GWP42004 and Placebo | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/12 | 0/13 | 0/12 | 1/14
Other Adverse Events (participants affected / at risk) | 7/11 | 8/12 | 11/13 | 11/12 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1:1 GWP42003 : GWP42004 (N=11) | 20:1 GWP42003 : GWP42004 (N=12) | GWP42003 and Placebo (N=13) | GWP42004 and Placebo (N=12) | Placebo (N=14)
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 | 0 | 0 | 0 — This event was added post study completion at the Sponsors request after review of the Beck Depression Inventory-II questionnaire responses.
Suicidal ideation (Psychiatric disorders) | 0 | 1 (1) | 0 | 0 | 0 — This event was added post study completion at the Sponsors request after review of the Beck Depression Inventory-II questionnaire responses.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1:1 GWP42003 : GWP42004 (N=11) | 20:1 GWP42003 : GWP42004 (N=12) | GWP42003 and Placebo (N=13) | GWP42004 and Placebo (N=12) | Placebo (N=14)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1
Vessel puncture site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Ear infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Genital candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 4 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW Pharmaceuticals Ltd (GW) will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.